CLINICAL TRIAL: NCT05436782
Title: Effects of Core Strengthening and Proprioceptive Neuromuscular Facilitation Pattern on Static Standing Balance and Plantar Pressure in Chronic Stroke
Brief Title: Effects of Core Strengthening and PNF Pattern on Balance and Plantar Pressure in Chronic Stroke
Acronym: PNF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/1089/2021
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Stroke; Paralysis
Keywords: Stroke, Static Balance, PNF, Plantar Pressure, PoData
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): • Group A (control group) will receive routine physical therapy involving muscle strengthening exercises, range of motion exercises, and stretching exercises up to the patient's tolerance. Other exercises will be pelvic bridging, rolling, sitting and standing exercises, walking practice and balancing in parallel bars, and wobble board exercises. Each session will be of 60 minutes 5 times weekly for 6 weeks
  Interventions: Other: Routine physical therapy
- Group B (Experimental): Group B (experimental group) will receive routine physical therapy for 20 minutes and additionally PNF technique (rhythmic initiation, and then agonistic reversals will be performed in lower extremity in D1 flexion pattern and D1 extension pattern up to patient's tolerance and core strengthening for 20 minutes 5 times weekly for 6 weeks. The outcome measure will be measured at and 6th week interval
  Interventions: Other: core strengthening exercises

INTERVENTIONS:
Other: core strengthening exercises — •Group B (experimental group) received routine physical therapy for 20 minutes and additionally PNF technique (rhythmic initiation, and then agonistic reversals were performed in the lower extremity in D1 flexion pattern and D1 extension pattern up to the patient's tolerance and core strengthening for 20 minutes 5 times weekly for 6 weeks. The outcome measure was measured at baseline and 6th-week interval
  Arms: Group B
Other: Routine physical therapy — •Group A (control group) will receive routine physical therapy involving muscle strengthening exercises, range of motion exercises, and stretching exercises up to the patient's tolerance. Other exercises were pelvic bridging, rolling, sitting and standing exercises, walking practice and balancing in parallel bars, and wobble board exercises. Each session was of 60 minutes 5 times weekly for 6 weeks
  Arms: Group A

SUMMARY:
To compare the effects of core strengthening and PNF on standing balance and plantar pressure in chronic stroke patients

DETAILED DESCRIPTION:
The effects of different exercise regimes and PNF techniques on balance and plantar pressure had been studied. This study focuses on determining the effects of CSE and PNF techniques on developing static standing balance and plantar pressure in stroke patients using PoData

ELIGIBILITY:
Inclusion Criteria:

* • Age 45-60

  * Score of 9 or higher on the static component of Berg Balance Scale
  * Both genders will be recruited.
  * First ever episode of stroke
  * Duration of stroke greater than 6 months.
  * Having a score of equal to or less than 2 on the Modified Ashworth Scale
  * Having a score of greater than or equal to 24 on the Mini-mental state examination in order to understand the commands.

Exclusion Criteria:

* • Concurrent orthopedic (for e.g. amputation ) that may hamper standing

  * Relevant psychiatric disorders that may prevent from following instructions.
  * Other medical drugs that may influence our intervention
  * Condition contraindicating physical activity
  * Use of cardiac pacemakers.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-14 (Estimated)

PRIMARY OUTCOMES:
Static Standing balance | 6 months
  It is measured using static component of berg balance scale. The items are scored from 0 to 4, with a score of 0 representing an inability to complete the task and a score of 4 representing independent item completion. Static component score is calculated out of 24 possible points. Scores of 0 to 9 represent static balance impairment, 10 to 15 represent acceptable static balance, and 15 to 24 represent good static balance

SECONDARY OUTCOMES:
Plantar pressure | 6 months
  PoData (Chinesport, Italy Version 5.0) this system provides information about weight distribution by measuring total body weight on fifth, first metatarsal and heel For a healthy individual the normal distribution is as follows 16.67% of the total body weight on the fifth metatarsal head, 33.33% of the total body weight on first metatarsal. 50% of the total body weight on heel

CONTACTS AND LOCATIONS:
Overall Officials: Sameed Liaqat, DPT, Principal Investigator — University of Lahore
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Punjqb, Pakistan

IPD SHARING:
Plan to Share IPD: No